CLINICAL TRIAL: NCT06411704
Title: Remote Exercise Video Adaptations to Maximize Physical Activity in Childhood Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REVAMP; NCI-2024-03931 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Frailty; Survivorship; Childhood Cancer
MeSH Terms: conditions — Frailty; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to leverage childhood cancer survivor input to adapt video content of a digital video disc-(DVD) delivered evidence-based PA intervention, originally designed for community-dwelling older adults.

Primary Objective:

- To leverage childhood cancer survivor input to adapt video content for an evidence-based remote exercise intervention.

DETAILED DESCRIPTION:
This study is being done to update existing exercise videos to suit adult survivors of childhood cancer to help them exercise at home. Patients will be asked to watch exercise videos designed for older adults and provide feedback during an interview to help researchers update the videos to childhood cancer survivors' preferences

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled in the St. Jude Lifetime Cohort (SJLIFE), aged 18- 39.
* Identifies as low active (self-reports <2 days/week of Physical Activity (PA) for at least 30 minutes over the past 6 months.
* Participant or legal guardian is able and willing to give informed consent.
* Internet access

Exclusion Criteria:

* Individuals who cannot speak, read, and/or understand English.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Long-term childhood cancer survivors with low physical activity.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Qualitative interviews | Day 1
  Semi-structured qualitative interviews will be utilized to collect participants' perspectives on relatability, functionality, and relevance of the exercise videos to childhood cancer survivors.
System Usability Scale Questionnaire | Day 1
  Multi-item Likert scored questionnaire to collect participants' perspectives on usability and relevance of the exercise videos. SUS scoring starts by calculating the sum of the score contributions from each item. Each item's score contribution will range from 0 to 4. For items 1,3,5,7,and 9 the score contribution is the scale position minus 1. For items 2,4,6,8 and 10, the contribution is 5 minus the scale position. Multiply the sum of the scores by 2.5 to obtain the overall value of SU. SUS scores have a range of 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Ness, PT, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols